CLINICAL TRIAL: NCT00340470
Title: Michigan Young Drivers Intervention Study
Brief Title: Michigan Driver Education Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 999903262; 03-CH-N262
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2007-02-06

CONDITIONS: Behavioral Intervention
Keywords: Injury; Motor Vehicle; Parenting; Randomized Trial; Behavioral Intervention
MeSH Terms: conditions — Wounds and Injuries

INTERVENTIONS:
Behavioral: Driver Education

SUMMARY:
Teens are at high risk for traffic violations and car crashes because of their young age, lack of driving experience, and exposure to high-risk driving conditions. The Checkpoints Program has used increased parental restrictions on teen driving through at least the first 4 months after their children obtain a driver's permit.

The purpose of this study is to evaluate the efficacy of the Checkpoints Program.

Approximately 400 teens in Michigan will participate in one of two study groups. One group will take standard driver education classes; the other group will take driver education classes that incorporate the Checkpoints Program. Teens and their parents will complete a written survey after completing the classes and a telephone survey after teens obtain a driver's permit. Teens will complete additional telephone surveys 1, 3, 6, and 12 months after obtaining a driver's permit. Researchers will use this information to study how parents manage teen driving practices, teen driving experiences (amount and conditions of), and high-risk teen driving behaviors.

DETAILED DESCRIPTION:
Teens are at high risk for traffic violations and motor vehicle crashes because of their young age, lack of driving experience, and exposure to high-risk driving conditions. Crash risk is greatest during the first two years of driving, and especially elevated during the first months of driving. Increasing parent involvement is becoming an important target of young driver education; however, little attention has been devoted to parental management of teen driving after teen licensure. Increased parental management of teen driving could reduce the risk of serious injury during the first months of driving and establish clear expectations for their teens' safe driving thereafter. In two randomized trials, the Checkpoints Program has been demonstrated to increase parental restrictions on teen driving through at least four months post-licensure. In this proposed research, we will evaluate the efficacy of the Checkpoints Program as applied to driver education. The purpose of this study is to assess the extent to which exposure to the Checkpoints Program during driver education classes in Michigan results in increased restrictions on young drivers during the first year of provisional licensure. The design is a randomized trial in which 24-30 commercial driver education classes will be randomly assigned to be either standard driver education or driver education that integrates the Checkpoints Program, Approximately 400 teens enrolled in driver education and one of their parents will be recruited and will complete written surveys at baseline and telephone surveys one month after teens obtained provisional licenses. Teens will complete additional telephone surveys one, three, six, and 12 months after provisional licensure. Study outcomes include parent management practices of teen driving, teen driving experience including the amount and conditions of driving during the first 12 months of licensure, and teen risky driving behaviors.

ELIGIBILITY:
* INCLUSION CRITERIA:

Teens between the ages of 15 years 0 months and 16 years 6 months enrolled in a licensed driver education course are eligible to participate.

EXCLUSION CRITERIA:

Adolescents over the age of 16 years 6 months or those whose parent or legal guardian does not attend the driver education course session to which they are specifically invited will be deemed ineligible for the study.

Ages: 15 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0
Dates: Start 2003-07-24; Study Completion 2007-02-06

PRIMARY OUTCOMES:
Adoption of the parent-teen driving agreement.

SECONDARY OUTCOMES:
Prent-imposed driving restrictions during the first 12 months of driving.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

REFERENCES:
- [Background] Doherty ST, Andrey JC, MacGregor C. The situational risks of young drivers: the influence of passengers, time of day and day of week on accident rates. Accid Anal Prev. 1998 Jan;30(1):45-52. doi: 10.1016/s0001-4575(97)00060-2. PMID 9542543